CLINICAL TRIAL: NCT03728699
Title: Microbiota Changes in Acute Myeloid Leukemia Patients Undergoing Intensive Chemotherapy
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2018NTLS107; HM2018-23 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sample Collection Blood — Collected from each patient twice weekly.
Diagnostic Test: Stool Sample — Collected from each patient twice weekly.

SUMMARY:
This is a prospective, observational study to collect stool and blood from acute myeloid leukemia patients undergoing intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 - 99 years) undergoing inpatient intensive chemotherapy for newly diagnosed, refractory, or relapsed AML. Patients may or may not have been exposed to any type of therapy before.
* Any intensive chemotherapy regimen defined as a planned ~4 week inpatient stay. Chemotherapy may be delivered for any number of days and on any schedule. Patients may be discharged from the hospital sooner than 4 weeks if the treating physician choose so, but the expectation at the initiation of chemotherapy must be ~4 weeks of inpatient stay, as is typical.
* Able to provide written voluntary consent before performance of any study related procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute myeloid leukemia (new diagnosis, refractory, or relapsed) undergoing any intensive chemotherapy with expected inpatient stay of ~4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Abundance of Phyla | Day 28
  Abundance in stool and circulating microbiota during intensive chemotherapy in patients with acute myeloid leukemia (AML), measured by16S rRNA gene profiling of biospecimens using the Illumina MiSeq platform
Abundance of Genera | Day 28
  Abundance in stool and circulating microbiota during intensive chemotherapy in patients with acute myeloid leukemia (AML), measured by16S rRNA gene profiling of biospecimens using the Illumina MiSeq platform

SECONDARY OUTCOMES:
Circulating Microbiota Diversity (Blood) | Day 28
  Describe circulating microbiota diversity over the course of treatment
Microbiota Diversity (Stool) | Day 28
  Describe stool microbiota diversity over the course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided